CLINICAL TRIAL: NCT05205551
Title: Prospera Test Evaluation in Cardiac Transplant (ProTECT)
Acronym: ProTECT
Status: Active, not recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-054-TRP
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Heart Transplant Rejection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ProTECT registry is an observational longitudinal, multi-center study observing patients undergoing heart transplant for whom Prospera testing is part of routine clinical care, who are enrolled within 60 days of heart transplantation.

DETAILED DESCRIPTION:
The ProTECT registry is an observational longitudinal, multi-center study observing patients undergoing heart transplant for whom Prospera™ testing is part of routine clinical care, who are enrolled within 60 days of heart transplantation. Patients who are enrolled in this study should have blood drawn for Prospera™ testing at regular intervals per routine clinical care. Prospera™ test results and results of surveillance endomyocardial biopsies, laboratory testing, echocardiograms, angiography and hemodynamic monitoring performed to monitor cardiac status and for signs of transplant rejection, as well as medications and post-transplant re-vascularization and surgical procedures will be recorded in the electronic case report form (eCRF). Patient management decisions, even those informed by the Prospera™ test result, are made based on the individual judgment of the healthcare providers participating in the study.

ELIGIBILITY:
Patients must meet all the following criteria to be eligible for the study:

1. Age 18 or older at the time of informed consent.
2. Enrolled within 60 days following heart transplantation.
3. Prospera™ testing is planned as part of standard clinical care to monitor for and assess transplant rejection.
4. Prospera™ testing is planned to be performed within 60 days (inclusive) following heart transplantation.
5. Selected by their healthcare provider to receive or continue receiving Prospera™ testing as part of their routine transplant management.
6. Willing and able to provide written informed consent.
7. Willing and able to comply with study procedures.

Patients are not eligible for the study if they meet any of the following criteria:

1. Pregnant at the time of signing informed consent.
2. Candidate for multiple solid organ or tissue transplant.
3. History of prior organ or cellular transplantation.
4. Ongoing testing with another allograft dd-cfDNA assessment is planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplantation Patients
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints: | 3 years
  Primary molecular endpoint: percent of donor-derived cell-free DNA (dd-cfDNA) measured via the Prospera™ test.
  Primary clinical endpoints:
  1. Biopsy-proven rejection (ISHLT Grade ACR >1R and ISHLT Grade AMR >0).
  2. Rejection with hemodynamic compromise (ejection fraction <40% or >20% decline from baseline or the need for inotropic agents in the absence of biopsy-proven rejection).
  3. Treated rejection (biopsy proven rejection or hemodynamic compromise rejection where immunosuppressive therapy was increased or augmented).

SECONDARY OUTCOMES:
Secondary Endpoints | 3 years
  The secondary endpoints are:
  1. The predictive performance of the Prospera™ test in detecting rejection or allograft dysfunction after heart transplant as measured by the sensitivity, specificity, negative predictive value, positive predictive value, and area under the curve (AUC) of the Prospera™ test
  2. Acute cellular rejection (ISHLT 2004 grade >1R)
  3. Antibody mediated rejection (ISHLT 2013 grade >0)
  4. Left ventricular ejection fraction (LVEF) measured by echocardiographic assessment
  5. Cardiac allograft vasculopathy (ISHLT grade >0)
  6. Cumulative mean fluorescence intensity (MFI) of donor specific antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Michael Olymbios, MD, Principal Investigator — Natera, Inc.
Locations (1):
- Natera, San Carlos, California, United States